CLINICAL TRIAL: NCT00674596
Title: The Effect of Renin Angiotensin System Blockage (RAS) Blockade On PTX3 Levels In Diabetic Patients With Proteinuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GATARAM2008
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes; Proteinuria; Renin Angiotensin System
Keywords: PTX3, ramipril, endothelial dysfunction; 1- Diabetic proteinuria; 2- The aim of this study was to find out whether the; beneficial effects of RAS blockage in diabetic; proteinuria has any relation with the alteration; of PTX3 levels.
MeSH Terms: conditions — Diabetes Mellitus; Proteinuria; Anterior segment mesenchymal dysgenesis | interventions — Ramipril

INTERVENTIONS:
Drug: ramipril — ramipril 10 mg/day during 3 months

SUMMARY:
Long pentraxin 3 (PTX3) is a recently discovered multimeric inflammatory mediator structurally linked to CRP and serum amyloid P-component. There is no data about the effects of Renin angiotensin system blockage (RAS) on PTX3 levels in diabetic patients with proteinuria. The aim of this study was to find out whether the beneficial effects of RAS blockage in diabetic proteinuria has any relation with the alteration of PTX3 levels. We searched for the effects of ACE inhibitor ramipril on the clinical and laboratory parameters of diabetic patients with proteinuria.

DETAILED DESCRIPTION:
The patients who were non-obese (BMI<30kg/m2), non dyslipidemic (total cholesterol <200mg/dl, Triglyceride<150mg/dl), and free of cardiovascular events (negative medical history, negative ECG findings) were investigated for enrollment. CKD stage 1 patients older than 18 years of age and willing to participate to the study were screened. From the 266 patients with established type 2 diabetes mellitus, 141 had proteinuria and/or hypertension (24 h protein excretion 1-2 g/day, systolic blood pressures ≥140mmHg and/or diastolic blood pressures ≥ 90 mmHg, respectively). All cases were first referrals and at the time of the study all were off treatment. Patients with history of coronary artery disease, smokers and those taking statins or renin-angiotensin blockers were excluded because of the effect of these factors on endothelial dysfunction. Of 141 screened patients 60 met the study criteria and were included in this study. The duration of proteinuria and diabetic nephropathy after initial diagnosis was not known.

The exclusion criteria were as follows: A)Nephrotic syndrome, B)coronary heart disease (patients with ischemic ST-T alterations and voltage criteria for LVH on electrocardiogram, and with history of revascularization or myocardial infarction), C) elevated liver enzymes (AST or ALT levels ≥ 40U/L) and D) renal failure (serum creatinine levels > 1.3 mg/dl).

In order to evaluate the effect of RAS blockade on plasma PTX3 concentrations, patients with proteinuria were given an ACE inhibitor (ramipril 5 mg/day) for 12 weeks. The effect of RAS blockade on insulin sensitivity and proteinuria was also investigated.

After the intervention period, blood samples were obtained for assay of plasma PTX3 concentrations, HbA1c , and insulin resistance scores (HOMA-IR). Urine samples were also collected over a 24-hour period to determine the degree of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 1 patients
* Older than 18 years of age
* Type 2 Diabetic patients
* Proteinuria

Exclusion Criteria:

* History of coronary artery disease
* Smokers
* Taking statins or renin-angiotensin blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-03; Study Completion 2008-03

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Yilmaz MI, Axelsson J, Sonmez A, Carrero JJ, Saglam M, Eyileten T, Caglar K, Kirkpantur A, Celik T, Oguz Y, Vural A, Yenicesu M, Lindholm B, Stenvinkel P. Effect of renin angiotensin system blockade on pentraxin 3 levels in type-2 diabetic patients with proteinuria. Clin J Am Soc Nephrol. 2009 Mar;4(3):535-41. doi: 10.2215/CJN.04330808. Epub 2009 Feb 11. PMID 19211665